CLINICAL TRIAL: NCT04166149
Title: Non-invasive Blood Test to Diagnose Acute Rejection After Pancreas and Kidney Transplantation: Pancreas and Renal Rejection Diagnosis Using Circulating Donor-derived Cell-free DNA in Peripheral Blood
Brief Title: Eliminating the Need for Pancreas Biopsy Using Peripheral Blood Cell-free DNA
Acronym: PancDX
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Wisconsin, Madison (Other); Georgetown University (Other)
Responsible Party: Principal Investigator, Jonathan Bromberg, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: Panc-DX
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Transplant;Failure,Kidney; Transplant; Failure, Pancreas; Rejection Acute Renal; Rejection Acute Pancreas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from recipients are taken in order to determine if peripheral blood has presence of donor-derived DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- University of Maryland: Pancreas and pancreas kidney patients enrolled at University of Maryland. Determine if dd-cfDNA exists in PTA, SPK, and PAK transplant recipient's blood by taking blood specimens at months 1-4, 6, 9, and 12 in the first year post transplant, and quarterly (month 15, 18, 21, 24) in the second year post transplant.
  Interventions: Diagnostic Test: dd-cfDNA Blood Test
- University of Wisconsin: Pancreas and pancreas kidney patients enrolled at University of Wisconsin. Determine if dd-cfDNA exists in PTA, SPK, and PAK transplant recipient's blood by taking blood specimens at months 1-4, 6, 9, and 12 in the first year post transplant, and quarterly (month 15, 18, 21, 24) in the second year post transplant.
  Interventions: Diagnostic Test: dd-cfDNA Blood Test
- Georgetown University: Pancreas and pancreas kidney patients enrolled at Georgetown University. Determine if dd-cfDNA exists in PTA, SPK, and PAK transplant recipient's blood by taking blood specimens at months 1-4, 6, 9, and 12 in the first year post transplant, and quarterly (month 15, 18, 21, 24) in the second year post transplant.
  Interventions: Diagnostic Test: dd-cfDNA Blood Test

INTERVENTIONS:
Diagnostic Test: dd-cfDNA Blood Test — The cfDNA measurement isolated from the peripheral blood contains small amounts from the graft. The blood sample is collected in Cell-Free DNA BCT (blood collection) tubes. These are measured by their difference in SNP (single nucleotide polymorphisms) genotype to determine the ratio of donor to recipient through shotgun sequencing. Higher levels of dd-cfDNA in a patient experiencing rejection is measured as a higher percentage of the total cf-DNA.

SUMMARY:
Donor-derived cell-free DNA (dd-cfDNA) has shown promise as an early marker for cellular injury caused by rejection. dd-cfDNA changes may also indicate other injuries that lead to progressive decline in transplant organ function associated with, in the case of kidney transplantation, the presence of interstitial fibrosis (IF) and tubular atrophy (TA) seen in biopsy specimens. Here, we will study the utility of dd-cfDNA to predict rejection in pancreas and pancreas-kidney recipients.

DETAILED DESCRIPTION:
+Objective The objective of this prospective observational study is to correlate circulating dd-cfDNA to clinical and sub-clinical acute rejection in pancreas transplant alone (PTA), pancreas after kidney (PAK), and simultaneous pancreas kidney (SPK) allograft recipients. The secondary objective study is to correlate circulating dd-cfDNA to pancreas and kidney function, using Hgb1c, C-peptide and insulin requirement to assess pancreas function, and using serum creatinine and estimated glomerular filtration rate (eGFR) to assess kidney function.

The clinical data and specimen collection will also enable future biomarker research.

+Study endpoints Serial dd-cfDNA in individuals over time will be correlated with clinical status and outcomes, such as events of allograft dysfunction or biopsy proven rejection.

The primary endpoints of the study are:

1. Clinical T cell as well as antibody mediated acute rejection
2. Sub-clinical T cell as well as antibody mediated acute rejection
3. Composite of clinical and sub-clinical T cell as well as antibody mediated acute rejection.

The secondary endpoints for the study are:

1. eGFR (estimated Glomerular Filtration Rate [mL/min]): will be derived from serum creatinine level, corrected for variables, using the CKD-RPI (Chronic Kidney Disease Epidemiology Collaboration) equation.
2. Renal allograft injury from BKV (Polyomaviridae polyomavirus) nephritis, CNI (calcineurin inhibitor) toxicity, acute pyelonephritis and recurrent disease confirmed by renal histology.
3. Pancreas allograft function derived from hemoglobin A1c, insulin requirement, and serum c-peptide per SOC
4. Pancreas allograft injury from pancreatitis (all causes, including gastrointestinal dysmotility or viral).
5. Correlate cfDNA levels with presence or absence of delayed graft function (DGF) and subsequent outcomes in a subset of enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult recipients (Age > 18 years )
2. All genders and all racial and ethnic groups
3. Pancreas transplant alone (PTA)
4. Simultaneous kidney-pancreas transplantation (SPK)
5. Pancreas-after-kidney (PAK) 6. Simultaneous pancreas and living donor kidney (SPLK)

7. Primary or re-transplants 8. Ability to come for follow-up and undergo biopsy (Performed in accordance to SOC) 9. Provided consent

Exclusion Criteria:

1. Pediatric recipients (Age < 18 years)
2. Pregnant women
3. Patients undergoing multi-organ transplants not otherwise specified (e.g., pancreas-liver, multi-visceral, or pancreas-heart)
4. Patients receiving donor kidney from an identical twin, as part of an SPLK (see above)
5. Did not provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with PTA, PAK, and SPK transplants. The data will compared to data obtained from the kidney transplant populations already investigated by CareDx in the DART and KOAR studies will be used as controls.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
dd-cfDNA correlation to acute rejection | August 1, 2019 to July 31, 2022
  To correlate circulating dd-cfDNA to clinical and sub-clinical acute rejection in PTA, PAK, and SPK allograft recipients.
  1. Clinical T cell as well as antibody mediated acute rejection.
  2. Sub-clinical T cell as well as antibody mediated acute rejection.
  3. Composite of clinical and sub-clinical T cell as well as antibody mediated acute rejection.

SECONDARY OUTCOMES:
dd-cfDNA correlation to pancreas and kidney function | August 1, 2019 to July 31, 2022
  To correlate circulating dd-cfDNA to pancreas and kidney function, using Hgb1c, C-peptide and insulin requirement to assess pancreas function, and using serum creatinine and estimated glomerular filtration rate [eGFR] to assess kidney function.
  1. eGFR (estimated Glomerular Filtration Rate [mL/min]): will be derived from serum creatinine level, corrected for variables, using the CKD-RPI (Chronic Kidney Disease Epidemiology Collaboration) equation.
  2. Renal allograft injury from BKV (Polyomaviridae polyomavirus) nephritis, CNI (calcineurin inhibitor) toxicity, acute pyelonephritis and recurrent disease confirmed by renal histology.
  3. Pancreas allograft function derived from hemoglobin A1c, insulin requirement, and serum C-peptide per SOC 4. Pancreas allograft injury from pancreatitis (all causes, including gastrointestinal dysmotility or viral).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - UW Health University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
As described in complete protocol.
Supporting Information: CSR
Time Frame: 2-3 years from study start.

REFERENCES:
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190
- [Background] Lo YM. Transplantation monitoring by plasma DNA sequencing. Clin Chem. 2011 Jul;57(7):941-2. doi: 10.1373/clinchem.2011.166686. No abstract available. PMID 21566070
- [Background] Snyder TM, Khush KK, Valantine HA, Quake SR. Universal noninvasive detection of solid organ transplant rejection. Proc Natl Acad Sci U S A. 2011 Apr 12;108(15):6229-34. doi: 10.1073/pnas.1013924108. Epub 2011 Mar 28. PMID 21444804
- [Background] Code of Federal Regulations, Title 42 - Public Health, Part 493 - Laboratory Requirements, Subpart A - General Provisions, Sections 1, 2 & 3.
- [Background] Streck, Cell-Free DNA BCT Instructions for Use: EXT-REF-Q-00002
- [Background] Hidestrand M, Tomita-Mitchell A, Hidestrand PM, Oliphant A, Goetsch M, Stamm K, Liang HL, Castleberry C, Benson DW, Stendahl G, Simpson PM, Berger S, Tweddell JS, Zangwill S, Mitchell ME. Highly sensitive noninvasive cardiac transplant rejection monitoring using targeted quantification of donor-specific cell-free deoxyribonucleic acid. J Am Coll Cardiol. 2014 Apr 1;63(12):1224-1226. doi: 10.1016/j.jacc.2013.09.029. Epub 2013 Oct 16. No abstract available. PMID 24140666
- [Background] Sigdel TK, Vitalone MJ, Tran TQ, Dai H, Hsieh SC, Salvatierra O, Sarwal MM. A rapid noninvasive assay for the detection of renal transplant injury. Transplantation. 2013 Jul 15;96(1):97-101. doi: 10.1097/TP.0b013e318295ee5a. PMID 23756769
- [Background] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192